CLINICAL TRIAL: NCT03748732
Title: Extensive Circumferential Partial Thickness Sclerectomy in Nanophthalmic Eyes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rafic Hariri University Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Mansour, MD, Clinical Professor, AUB, Professor, Rafic Hariri University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RaficHaririUHAMM
Record Dates: First submitted 2018-11-18; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Nanophthalmos
Keywords: uveal effusion
MeSH Terms: conditions — Microphthalmos

STUDY DESIGN:
Intervention Model Description: surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: sclerectomy — scleral flap
  Other Names: maximal scleral excision

SUMMARY:
Purpose: To describe an extensive scleral excision technique to treat or prevent uveal effusion in nanophthalmic eyes.

Design: Prospective interventional case series.

Methods:

* Setting: Institutional.
* Patient Population: Consecutive patients with nanophthalmos were operated on by one surgeon.
* Intervention Procedure: A single, 90% thickness scleral window extending from immediately behind the extraocular muscle insertions to the vortex veins was performed for 3 and 1/4 quadrants as a circumferential strip.
* Main Outcome Measure: Resolution or prevention of uveal effusion.

DETAILED DESCRIPTION:
Surgical Technique All surgeries were performed under general anesthesia by one surgeon (AMM). Because the majority of the patients were young with narrow palpebral fissures and very deep set globes in small orbits, special surgical techniques were required. Lateral canthotomy was performed on all patients except for the first. Limbal 360o conjunctival peritomy was followed by securing of each rectus muscles with a modified muscle hook and 2-0 silk suture. Scleral dissection was performed from immediately behind to the muscle insertions posterior to the vortex veins. A 90% depth scleral window was excised over 3 and ¼ quadrants, excluding 3/4 of the superior temporal quadrant to avoid damaging the superior oblique muscle.

ELIGIBILITY:
Inclusion Criteria: nanophthalmos -

Exclusion Criteria: None

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
resolution of uveal effusion | 1 month
  disappearence of uveal effusion by OCT

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Mansour, MD, Study Chair — Rafic Hariri University Hospital
Locations (1):
- Rafic Hariri University Hospital, Beirut, South Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided
if part of collaboration, we will share the data

REFERENCES:
- [Result] Carricondo PC, Andrade T, Prasov L, Ayres BM, Moroi SE. Nanophthalmos: A Review of the Clinical Spectrum and Genetics. J Ophthalmol. 2018 May 9;2018:2735465. doi: 10.1155/2018/2735465. eCollection 2018. PMID 29862063
- [Derived] Mansour A, Stewart MW, Shields CL, Hamam R, Abdul Fattah M, Sheheitli H, Mehanna CJ, Yassine S, Chahine H, Keaik M, Maalouf F, Jaroudi M. Extensive circumferential partial-thickness sclerectomy in eyes with extreme nanophthalmos and spontaneous uveal effusion. Br J Ophthalmol. 2019 Dec;103(12):1862-1867. doi: 10.1136/bjophthalmol-2018-313702. Epub 2019 Mar 15. PMID 30877130